CLINICAL TRIAL: NCT02794311
Title: AlcoholPredict: Neuropsychology, Brain Imaging and Genetic Polymorphisms in Binge Drinking
Brief Title: Risk Factors Associated With Binge Drinking Behaviors Among College Students
Acronym: AlcoolPredict
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PO13129
Record Dates: First submitted 2016-05-12; First posted 2016-06-09 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2020-06

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Alcoolpredict — psychological (personality), neuropsychological (executive functions, memory), genetic (snp polymorphisms) and neuro-anatomical (fMRI)

SUMMARY:
The purpose of this study is to specify the psychological, cognitive, neuro-functional and genetic profile associated with binge drinker behaviors among young adults. Results will help identifying more precisely vulnerability factors associated with this pattern of alcohol consumption and guiding prevention efforts.

DETAILED DESCRIPTION:
Binge drinking behavior is characterised by speed of drinking on a particular occasion, frequency of drunkenness during the most recent six month period, and the percentage of times getting drunk when drinking. The prevalence of weekly binge drinking among European Union drinkers in 2009 was reported to be 28% of the student population, and 33% among all young people aged 15-24. The consequences of this behavior are multiple and often dramatic, they include: academic failure, violent acts, rape, domestic or road accidents. The study aims to identify vulnerability factors associated with binge drinking. The protocol explores the psychological (personality), neuropsychological (executive functions, memory), genetic (snp polymorphisms) and neuro-anatomical (fMRI) patterns associated with binge drinking behavior.

ELIGIBILITY:
Inclusion criteria :

* Males or females
* Right-handed
* Aged 18-25 years
* Native French speaker, able to read French and complete study evaluations
* Caucasian
* Able to provide informed written and verbal consent

Exclusion criteria

* A significant general medical illness, including neurological disorders, mental retardation or head trauma
* Depression, bipolar disorder, schizophrenia or schizoaffective disorder diagnostic according to DSM-IV
* Handling of psychotropics substances
* A sensorial impairment (visual and/or hearing)
* Women who are pregnant
* Contraindication to the use of MRI (pacemaker, metal in their body)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2015-02; Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test : Mini International Neuropsychiatric Interview (M.I.N.I) | day 1
Neuropsychological test : Wisconsin Card Sorting Test (WCST) | V2(3 weeks later)
Genetics tests (Single Nucleotide Polymorphism) | V2(3 weeks later)
MRI - signal BOLD (" Blood Oxygen Level Dependant "). | V3(up to 2 month)
Neuropsychological test : Family Informant Schedule and Criteria (FISC) | day 1
Neuropsychological test : Alcohol Use Questionnaire | day 1
Neuropsychological test :Trail Making Test, partie A et B | V3(up to 2 month)
Neuropsychological test : Plus/Minus Test | V3(up to 2 month)
Neuropsychological test :Go/No-Go | V3(up to 2 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Result] Lannoy S, Dricot L, Benzerouk F, Portefaix C, Barriere S, Quaglino V, Naassila M, Kaladjian A, Gierski F. Neural Responses to the Implicit Processing of Emotional Facial Expressions in Binge Drinking. Alcohol Alcohol. 2021 Feb 24;56(2):166-174. doi: 10.1093/alcalc/agaa093. PMID 33075804